CLINICAL TRIAL: NCT01216527
Title: A Phase III, Multicenter Randomized Controlled Study of Neo-adjuvant Chemoradiotherapy Followed by Surgery Versus Surgery for Locally Advanced Squamous Cell Esophageal Carcinoma
Brief Title: Phase III Study of Neo-adjuvant Chemoradiotherapy Followed by Surgery for Squamous Cell Esophageal Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: Affiliated Cancer Hospital of Shantou University Medical College (Other); Shanghai Chest Hospital (Other); Fudan University (Other); Zhejiang Cancer Hospital (Other); Taizhou Hospital (Other); The Second People's Hospital of Sichuan (Other); Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Principal Investigator, Jianhua Fu, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2007048
Record Dates: First submitted 2010-10-06; First posted 2010-10-07 (Estimated); Last update posted 2017-02-27 (Actual); Status verified 2017-02

CONDITIONS: Squamous Cell Esophageal Carcinoma
Keywords: Stage IIB or III squamous cell esophageal carcinoma.
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- experimental group (Experimental): Neo-adjuvant Chemoradiotherapy followed by Surgery
  Interventions: Procedure: Neo-adjuvant Chemoradiotherapy followed by Surgery
- control group (Active Comparator): only Surgery
  Interventions: Procedure: surgery

INTERVENTIONS:
Procedure: Neo-adjuvant Chemoradiotherapy followed by Surgery — 1. Radiotherapy combined with concomitant chemotherapy:
     Radiotherapy Program:External radiation with a total dose of 40.0Gy is given in 20 fractions of 2.0Gy,5 fractions a week.
     neo-chemotherapy program: Vinorelbine 25mg/m2, IV (in the vein) on day 1 and day 8 of each 21 day cycle. Cisplatin 75mg/m2,IV DRIP on day 1 of each 21 day cycle;or Cisplatin 25mg/m2,IV DRIP on day 1 to day 4 of each 21 day cycle.
     Number of cycles:two
  2. surgery:Mckeown Modification Surgery and total two-field lymphadenectomy
  Arms: experimental group
Procedure: surgery — two field lymphadenectomy
  Arms: control group

SUMMARY:
The primary objective is to compare neo-adjuvant chemoradiotherapy followed by surgery versus surgery, in terms of the overall survival time (OS) in patients with Stage IIB or III squamous cell esophageal carcinoma.

DETAILED DESCRIPTION:
Esophageal cancer (EC) is the eighth most common cancers in the world, with more than 480,000 new cases and 400,000 deaths occurred annually worldwide. In China, every year, no matter new cases or deaths account for more than half of the world. Besides, over 90% of Chinese patients have esophageal squamous cell carcinoma (ESCC).

Surgery is the main treatment of this disease, but the prognosis of patients with locally advanced esophageal cancer is rather poor. As a result of surgery alone, the 5-year survival rate of about 25% has not changed significantly in several decades.

Preoperative chemoradiotherapy followed by surgery seems to hopefully improve the survival of EC. Nevertheless, the results of different studies were inconsistent. Recently, the CROSS trial has demonstrated that preoperative chemoradiotherapy can significantly increased the overall survival of patients with EC compared with surgery alone. It should be noticed that only 84 cases(23%) of ESCC were enrolled in this trial with potential minimal follow-up of 2 years, which may be not perfect to evaluate the effect of this combined therapy for this tumor type.

Up till now, vinorelbine has no indications for esophageal cancer, although, some studied have reported its effect and feasibility to the therapy of EC. Vinorelbine has similar mechanism with paclitaxel and docetaxel, which are recommended for the chemotherapy of EC by NCCN. They are all classified as antimicrotubule agents, which cause mitotic arrest and eventual cell death through inhibition of microtubule dynamics. In comparison with the taxanes, vinorelbine has obvious advantage of few cardiac toxicity. This should be beneficial to prevent cardiac side effects of chemoradiotherapy, especially for the middle or lower thoracic EC, which account for over 70% of thoracic EC in China. For this group of patients, radiotherapy can hardly avoid cardiac toxicity.

Based on our preliminary study, we have demonstrated the validity and safety of vinorelbine and cisplatin-based neoadjuvant chemoradiotherapy.

We are to carry out a phased III clinical trial to investigate the effect of this multidisciplinary therapy for the overall survival of patients with locally advanced ESCC.

ELIGIBILITY:
Inclusion Criteria:

1. Histologic diagnosis of squamous cell thoracic esophageal carcinoma of Stage IIB or III, which is potentially resectable.
2. Patients must not have received any prior anticancer therapy.
3. More than 6 months of expected survival.
4. Age ranges from 18 to 70 years.
5. Absolute white blood cells count ≥4.0×109/L, neutrophil ≥1.5×109/L, platelets ≥100.0×109/L, hemoglobin ≥90g/L, and normal functions of liver and kidney.
6. Karnofsky performance status (KPS) of 90 or more.
7. Signed informed consent document on file.

Exclusion Criteria:

1. Patients are diagnosed or suspected to be allergic to cisplatin or vinorelbine.
2. Patients with concomitant hemorrhagic disease.
3. Pregnant or breast feeding.
4. Inability to use gastric conduit after esophagectomy because of a prior surgery.
5. Patients with concomitant peripheral neuropathy, whose CTC status is 2 or even more.
6. Have a prior malignancy other than esophageal carcinoma, carcinoma in situ of the cervix, nonmelanoma skin cancer or cured early stage of prostate cancer.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 430 (Estimated)
Dates: Start 2007-06; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Overall survival rate | 3 and 5 years

SECONDARY OUTCOMES:
toxicities of neo-adjuvant chemoradiotherapy | 56 days
  Evaluate the toxicities of neo-adjuvant chemoradiotherapy,according to National Cancer Institute Common Terminology Criteria for Adverse Event,Version 3.0(CTC AE3.0).
assessment in perioperation | perioperative period
  Removal rate， Time of operation， Quantity of bleeding， Thoracic Drainage， Days of Hospitalization， Rate of Operative Complication， Mortality of perioperation，
efficacy of neo-adjuvant chemoradiotherapy | 4 weeks after completion of radiotherapy
  Criteria:Response Evaluation Criteria in Solid Tumors，RECIST
Disease free survival rate | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Jian-hua Fu, Professor, Principal Investigator — Sun Yat-sen University
Locations (2):
- China (2):
  - Sun Yat-sen Uniersity Cancer Center, Guangzhou, Guangdong
  - Cancer Hospital of Shantou University Medical College, Shantou, Guangdong

REFERENCES:
- [Background] Jemal A, Bray F, Center MM, Ferlay J, Ward E, Forman D. Global cancer statistics. CA Cancer J Clin. 2011 Mar-Apr;61(2):69-90. doi: 10.3322/caac.20107. Epub 2011 Feb 4. PMID 21296855
- [Background] Herskovic A, Russell W, Liptay M, Fidler MJ, Al-Sarraf M. Esophageal carcinoma advances in treatment results for locally advanced disease: review. Ann Oncol. 2012 May;23(5):1095-1103. doi: 10.1093/annonc/mdr433. Epub 2011 Oct 14. PMID 22003242
- [Background] van Hagen P, Hulshof MC, van Lanschot JJ, Steyerberg EW, van Berge Henegouwen MI, Wijnhoven BP, Richel DJ, Nieuwenhuijzen GA, Hospers GA, Bonenkamp JJ, Cuesta MA, Blaisse RJ, Busch OR, ten Kate FJ, Creemers GJ, Punt CJ, Plukker JT, Verheul HM, Spillenaar Bilgen EJ, van Dekken H, van der Sangen MJ, Rozema T, Biermann K, Beukema JC, Piet AH, van Rij CM, Reinders JG, Tilanus HW, van der Gaast A; CROSS Group. Preoperative chemoradiotherapy for esophageal or junctional cancer. N Engl J Med. 2012 May 31;366(22):2074-84. doi: 10.1056/NEJMoa1112088. PMID 22646630
- [Background] Kulke MH, Muzikansky A, Clark J, Enzinger PC, Fidias P, Kinsella K, Michelini A, Fuchs CS. A Phase II trial of vinorelbine in patients with advanced gastroesophageal adenocarcinoma. Cancer Invest. 2006 Jun-Jul;24(4):346-50. doi: 10.1080/07357900600705268. PMID 16777685
- [Background] Airoldi M, Cortesina G, Giordano C, Pedani F, Bumma C, Gabriele P. Docetaxel and vinorelbine: an effective regimen in recurrent squamous cell esophageal carcinoma. Med Oncol. 2003;20(1):19-24. doi: 10.1385/MO:20:1:19. PMID 12665680
- [Background] Koussis H, Scola A, Bergamo F, Tonello S, Basso U, Karahontzitis P, Chiarion-Sileni V, Pasetto L, Ruol A, Loreggian L, Lora O, Bottin R, Marioni G, Donach M, Jirillo A. Neoadjuvant carboplatin and vinorelbine followed by chemoradiotherapy in locally advanced head and neck or oesophageal squamous cell carcinoma: a phase II study in elderly patients or patients with poor performance status. Anticancer Res. 2008 Mar-Apr;28(2B):1383-8. PMID 18505084
- [Background] Yang H, Fu JH, Hu Y, Lin P, Liu MZ, Li Q, Fang ZC, Hu YH. [Neo-adjuvant chemoradiotherapy followed by surgery in treatment of advanced esophageal carcinoma]. Zhonghua Yi Xue Za Zhi. 2008 Dec 9;88(45):3182-5. Chinese. PMID 19171088
- [Derived] Yang H, Liu H, Chen Y, Zhu C, Fang W, Yu Z, Mao W, Xiang J, Han Y, Chen Z, Yang H, Wang J, Pang Q, Zheng X, Yang H, Li T, Zhang X, Li Q, Wang G, Chen B, Mao T, Kong M, Guo X, Lin T, Liu M, Fu J. Long-term Efficacy of Neoadjuvant Chemoradiotherapy Plus Surgery for the Treatment of Locally Advanced Esophageal Squamous Cell Carcinoma: The NEOCRTEC5010 Randomized Clinical Trial. JAMA Surg. 2021 Aug 1;156(8):721-729. doi: 10.1001/jamasurg.2021.2373. PMID 34160577
- [Derived] Liu S, Wen J, Yang H, Li Q, Chen Y, Zhu C, Fang W, Yu Z, Mao W, Xiang J, Han Y, Zhao L, Liu H, Hu Y, Liu M, Fu J, Xi M. Recurrence patterns after neoadjuvant chemoradiotherapy compared with surgery alone in oesophageal squamous cell carcinoma: results from the multicenter phase III trial NEOCRTEC5010. Eur J Cancer. 2020 Oct;138:113-121. doi: 10.1016/j.ejca.2020.08.002. Epub 2020 Aug 30. PMID 32877795
- [Derived] Yang H, Liu H, Chen Y, Zhu C, Fang W, Yu Z, Mao W, Xiang J, Han Y, Chen Z, Yang H, Wang J, Pang Q, Zheng X, Yang H, Li T, Lordick F, D'Journo XB, Cerfolio RJ, Korst RJ, Novoa NM, Swanson SJ, Brunelli A, Ismail M, Fernando HC, Zhang X, Li Q, Wang G, Chen B, Mao T, Kong M, Guo X, Lin T, Liu M, Fu J; AME Thoracic Surgery Collaborative Group. Neoadjuvant Chemoradiotherapy Followed by Surgery Versus Surgery Alone for Locally Advanced Squamous Cell Carcinoma of the Esophagus (NEOCRTEC5010): A Phase III Multicenter, Randomized, Open-Label Clinical Trial. J Clin Oncol. 2018 Sep 20;36(27):2796-2803. doi: 10.1200/JCO.2018.79.1483. Epub 2018 Aug 8. PMID 30089078
- [Derived] Wen J, Yang H, Liu MZ, Luo KJ, Liu H, Hu Y, Zhang X, Lai RC, Lin T, Wang HY, Fu JH. Gene expression analysis of pretreatment biopsies predicts the pathological response of esophageal squamous cell carcinomas to neo-chemoradiotherapy. Ann Oncol. 2014 Sep;25(9):1769-1774. doi: 10.1093/annonc/mdu201. Epub 2014 Jun 6. PMID 24907633